CLINICAL TRIAL: NCT05333588
Title: The Safety and Efficacy Study of Autologous Tumor-infiltrating Lymphocyte (TILs) Therapy Combined With Conventional Chemotherapy for Patients With Advanced Stage of Glioblastoma Multiforme.
Brief Title: The Safety Study of Autologous TILs Therapy for Patients With Glioblastoma Multiforme.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Senlang Biotechnology Inc., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TILs for Glioblastoma
Record Dates: First submitted 2022-04-01; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Glioblastoma Multiforme, Adult
Keywords: glioma; TiLs; Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tumor infiltrating lymphocyte (Experimental): 1x10^9-5x10^10 of autologous TILs will be adoptive transfer to patients.
  Interventions: Biological: Tumor Infiltrating Lymphocytes (TIL)

INTERVENTIONS:
Biological: Tumor Infiltrating Lymphocytes (TIL) — The autologous TILs will be intravenous infused into patients.
  Other Names: TILs

SUMMARY:
The study is to evaluate the safety and efficacy of tumor infiltrating lymphocyte (TIL) therapy for patients with maligant glioblastoma multiforme. Autologous TiLs should be given by intravenous infusion after 5 days of lymphodepletion treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 80 years old;
2. Has at least one measurable tumor foci;
3. ECOG score range : 0-2;
4. Expected survival time: ≥ 3 months;
5. All screening labs should be performed 7 days prior to registration.The laboratory results need to meet below criteria:

   * Absolute white blood cell counts (WBC) ≥ 3.0×10^9/L；
   * Platelet count (PLT) ≥ 100×10^9/L；
   * Hematological Absolute neutrophil count (ANC) ≥ 1.5×10^9/L；
   * Hemoglobin (HGB) ≥ 90g/L;
   * Albumin (absolute) ≥ 2.8g/dL;
   * Serum ALT/AST ≤ 2.5×ULN (for patients with liver metastasis ≤ 5×ULN);
   * Total bilirubin (TBIL) ≤ 1.5×ULN (for patients with liver metastasis ≤ 2×ULN);
   * Renal Serum creatinine OR measured or calculated a creatinine clearance (CR) ≤1.5×ULN OR≥ 50 mL/min for participant;
   * AST/ALT (SGOT) ≤ 2.5×ULN (for patients with liver metastasis ≤ 5×ULN);
   * International Normalized Ratio (INR) ≤ 1.5;
   * Prothrombin Time (PT) and Activated Partial Thromboplastin Time (APTT) ≤ 1.5×ULN;
6. Female participant of childbearing potential should have a negative result of human chorionic gonadotropin (HCG) test. The participants must take contraception during the entire clinical follow-up.
7. Be willing and able to provide written informed consent/assent for the trial.

Exclusion Criteria:

1. Has systemic active infection and requiring treatment;
2. Has severe physical or mental illness;
3. Has active rheumatic disease;
4. Has any kinds of organ transplantation;
5. Being pregnant or lactating;
6. Enrolled in other clinical trials within 4 weeks prior to registration;
7. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies), active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C;
8. Other conditions that the researcher considered to be excluded;
9. Has taken blow treatment before enrollment:

   * Received systemic immunosuppressive treatments, aside from corticosteroids within 14 days of treatment;
   * Plan to get inactivated vaccine 28 days prior/during, or 60 days post the treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events related to TiLs infusion | 1 month
  The primary outcome measure of this clinical trial is accessed by the safety of the TILs product. The safety profile for TILs is characterized by its incidence of the adverse events.

SECONDARY OUTCOMES:
Progressional free of survival (PFS) | Up to 24 months
  PFS is defined as the duration of time from start of treatment to time of progression. All patients will be followed for a minimum of 2 years.
Objective response rate (ORR) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Chunyan Li, academician, Principal Investigator — Member of the Chinese Academy of Engineering
Locations (1):
- The Second Hospital of HeBei Medical University, Shijiazhuang, Hebei, China